CLINICAL TRIAL: NCT00897910
Title: Strategies to Isolate and Expand Myeloma Specific T-cells Using Autologous B Cells as Antigen Presenting Cell B-APC
Brief Title: Studying T Cells in Blood and Bone Marrow Samples From Patients With Multiple Myeloma
Status: Terminated | Type: Observational
Why Stopped: Funding unavailable
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Zaid Al-Kadhimi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Other Study IDs: CDR0000597015; P30CA022453 (NIH); WSU-2007-070
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Results first posted 2013-12-12 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Flow Cytometry; Immunoenzyme Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Data from flow cytometry, and Cytokine release assays for B cells and T cells from peripheral blood mononuclear cells (PBMCs) will be obtained.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: flow cytometry — Collection of PBMCs over a period of 9-12 months, and the laboratory component will be performed over another year.
Other: immunoenzyme technique — Collection of PBMCs over a period of 9-12 months, and the laboratory component will be performed over another year.
Other: laboratory biomarker analysis — Collection of PBMCs over a period of 9-12 months, and the laboratory component will be performed over another year.

SUMMARY:
RATIONALE: Studying samples of blood and bone marrow from patients with cancer in the laboratory may help doctors learn more about T cells and plan better treatment for multiple myeloma.

PURPOSE: This research study is looking at T cells in blood and bone marrow samples from patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the feasibility of expanding myeloma-specific T cells using autologous ex vivo expanded B cells loaded with myeloma antigens as antigen-presenting cells (B-APCs) in peripheral blood and bone marrow samples from patients with multiple myeloma.

Secondary

* To examine the feasibility of selecting and expanding myeloma-specific T cells ex vivo using interferon γ release and CD3/CD28 stimulation.

OUTLINE: Peripheral blood and bone marrow samples are collected periodically for laboratory studies. Samples are analyzed to assess the feasibility of expanding autologous B cells ex vivo using CD40L and IL-4; the antigen-presenting phenotype of autologous B-cell antigen-presenting cells (B-APCs) using flow cytometry; and the antigen-presenting function of B-APCs using ELISPOT and chromium-release assay. Myeloma-specific interferon γ secreting T cells are isolated and selected using Miltenyi beads. The selected myeloma-specific T cells are expanded ex vivo using anti CD3/CD28 beads.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of multiple myeloma identified from the outpatient clinics or inpatient service of Karmanos Cancer Center by physicians in the Department of Hematology and Medical Oncology.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Al-Kadhimi, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the outpatient clinics or inpatient service of Karmanos Cancer Center by physicians in the Department of Hematology and Medical Oncology, between April 2008 and October 2009.
Pre-assignment Details: All 6 consented subjects had blood drawn during their routine labs. No bone marrow samples were collected.
Period: Overall Study
Arm/Group | Collection of Circulating Blood and Bone Marrow.
Started | 6 (None of the blood samples were analyzed due to lack of funding. No tissue sample was collected.)
Completed | 6 (None of the blood samples were analyzed due to lack of funding. No tissue sample was collected)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Collection of Circulating Blood and Bone Marrow.
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Myeloma-specific T Cells ex Vivo Expanded Using Flow Cytometry
Time Frame: Collection of PBMCs over a period of 9-12 months, and the laboratory component will be performed over another year.
Arm/Group | Collection of Blood and Bone Marrow.
Number analyzed (Participants) | 0

2. Secondary Outcome: Cell Counts of Myeloma-specific T Cells ex Vivo Expanded Before and After CD3/CD28 Stimulation
Time Frame: Collection of PBMCs over a period of 9-12 months, and the laboratory component will be performed over another year.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Collection of Circulating Blood and Bone Marrow.
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Tis study was closed due to technical laboratory difficulty in performing the experiments proposed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes